CLINICAL TRIAL: NCT06854224
Title: Orexin Antagonism to Target Mechanisms of Suicide Risk: A Proof-of-Concept Clinical Trial
Brief Title: Orexin Antagonism for Suicide Risk: A Proof-of-Concept Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marianne Goodman (Other)
Collaborators: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Marianne Goodman, Psychiatrist; VISN 2 MIRECC Director, Bronx Veterans Medical Research Foundation, Inc
Organization: Bronx Veterans Medical Research Foundation, Inc (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1851192
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Suicide Risk; Major Depressive Disorder (MDD)
Keywords: Suicide risk; Proof-of-concept clinical trial; Suvorexant; Orexin antagonist
MeSH Terms: conditions — Depressive Disorder, Major | interventions — suvorexant; Orexin Receptor Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Suvorexant group (Experimental): Veteran patients with Major Depressive Disorder and elevated risk of suicide will receive the FDA-approved drug Suvorexant (brand name: Belsomra), a mixed Orexin antagonist, for four weeks. Participants will take 10mg of Surovexant nightly for the first two weeks and 20mg of Surovexant nightly for the second two weeks.
  Interventions: Drug: Suvorexant (dual orexin receptor antagonist)

INTERVENTIONS:
Drug: Suvorexant (dual orexin receptor antagonist) — Veteran patients with Major Depressive Disorder and elevated risk of suicide will receive the FDA-approved drug Suvorexant (brand name: Belsomra), a dual orexin receptor antagonist, for four weeks. Participants will take 10mg of Surovexant nightly for the first two weeks and 20mg of Surovexant nightly for the second two weeks.

SUMMARY:
The goal of this proof-of-concept clinical trial is to evaluate the initial safety, feasibility, and tolerability of the orexin mixed antagonist suvorexant in a sample of veteran adults with Major Depressive Disorder and elevated suicide risk. The main question it aims to answer is: Is Suvorexant safe, feasible, and tolerable for participants?

Participants will:

* Take Surovexant every day for four weeks (10mg in the first two weeks and 20mg in the second two weeks)
* Visit the medical center at the beginning of the study (week 1), after taking Suvorexant for two weeks (week 3) and following the full Suvorexant dose (week 5) for in-person assessments.
* Fill out self-report assessments (remotely) at week 2 (after one week of Suvorexant) and week 4 (after three weeks of Surovexant)

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* At least 18 years of age (up to 70 years)
* Primary diagnosis of Major Depressive Disorder as determined by the study psychiatrist and confirmed by the Mini-International Neuropsychiatric Interview (MINI)
* Lifetime suicide attempt history and suicidal ideation at baseline as determined by a score ≥2 on the Columbia-Suicide Severity Rating Scale (C-SSRS)

Exclusion Criteria:

* Clinically significant medical or neurological condition
* Current use of strong CYP3A live enzymes or moderate CYP3A inhibitors or strong CYP3A inducers
* Current use of digoxin
* Currently pregnant, not using contraception, nursing, or trying to become pregnant
* Active substance use disorder in the last six months, disorder, or current or past psychotic disorder, bipolar disorder, or obsessive-compulsive disorder
* Severe traumatic brain injury
* Imminent suicidal or homicidal risk
* Free of unstable medical conditions or any contraindication to suvorexant (per FDA prescribing label) as determined by patient interview and review of available medical records.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Implicit Association Tests (IATs) | Weeks 1, 3, and 5
  Implicit Association Tests ( IATs) use reaction time (RT) to capture automatic, implicit processes to gauge implicit self-identification with a construct of interest. Participants classify stimuli presented in the center of the screen into categories. The category labels are located on the left and right of the screen and participants classify stimuli by selecting keys corresponding to the left or right. RTs are measured as participants complete this task thereby gauging implicit mental associations. This study uses two variations of the IAT, a suicide-related IAT and a Escape-Me IAT to determine the extent to which participants associate suicide-related and escape-related constructs with the self.

SECONDARY OUTCOMES:
Buss-Perry Aggression Questionnaire | Weeks 1, 2, 3, 4, and 5
  The Buss-Perry Aggression Questionnaire is a 20-item self-report questionnaire assessing four dimensions of aggression: physical aggression, verbal aggression, anger, and hostility. Participants indicate how well each item describes them on a 5-point scale ranging from 1 (Not at all like me) to 5 (Very much like me).
Overt Aggression Scale Modified | Weeks 1, 2, 3, 4, and 5
  The Overt Aggression Scale Modified (OAS-M) is a clinician-administered interview of aggressive behavior. Participants are asked about "outbursts of anger" (reactive aggression) in the past week. The OAS-M is strongly related to measures of anger and differentiates between participants with and without intermittent explosive disorder, supporting its validity as a measure of reactive aggression.
Point Subtraction Aggression Paradigm | Weeks 1, 3, and 5
  The Point Subtraction Aggression Paradigm (PSAP) is a laboratory-based assessment of reactive aggression in which participants play a competitive computer game against a fictional opponent to obtain points that coincide with a monetary reward. The PSAP can be administered virtually through Inquisit Web, a software designed to facilitate virtual research experiments.
Barratt Impulsiveness Scale | Weeks 1, 2, 3, 4, and 5
  The Barratt Impulsiveness Scale (BIS-11) is a 30-item self-report questionnaire assessing the personality/behavioral construct of impulsiveness. It includes six first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and three second-order factors (attentional, motor, and non-planning impulsiveness). Participants rate each item on a 4-point scale ranging from 1 (Rarely/Never) to 4 (Almost Always/Always). Total scores can range from 30 to 120.
Beck Scale for Suicidal Ideation | Weeks 1, 2, 3, 4, and 5
  The Beck Scale for Suicidal Ideation (BSSI) is a 21-item self-report questionnaire assessing suicidal thinking that helps identify individuals at risk. It also measures a broad spectrum of suicide-related attitudes and behaviors. The first five items are often used as the screener, where participants are directed to item 20 if they score 0 on these items. The overall score is computed by totaling up the scores on the first 19 items. Each item is rated from 0 to 2. Scores range from 0 to 38, with a higher score indicating a higher level of suicide ideation.
Columbia Suicide Severity Rating Scale | Weeks 1, 2, 3, 4, and 5
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a clinician-administered questionnaire assessing suicidal ideation and behavior with four subscales: ideation severity (five types of ideation of increasing severity), intensity of ideation (Frequency, Duration, Controllability, Deterrents, and Reasons for Ideation), suicidal behavior (4 types of suicidal behaviors - actual, interrupted, aborted attempts and preparatory behaviors - and the total number), and behavior lethality (For suicide attempts or non-suicidal self-injurious behavior).
Gradual-Onset Continuous Performance Task | Weeks 1, 3, 5
  The gradCPT task is a continuous performance task designed to measure sustained attention and response inhibition. It involves monitoring a continuous stream of natural scenes from two categories-cities and mountains-with a 9:1 ratio. Participants respond either to the frequent or rare category, yielding a response rate of either 90% or 10%. The task is associated with substantial and stable individual differences, with performance correlating significantly with network connectivity both during task performance and in resting states. The gradCPT task is an important new paradigm in attention research, providing insights into the neural network of sustained attention and the role of response inhibition in performance.
Emotional Gradual Onset Continuous Performance Task | Weeks 1, 3, and 5
  The Emotional Gradual Onset Continuous Performance Task (emogradCPT), is used to characterize the impact of emotional distractors (background images) on the ability to sustain attention during an emotionally neutral task (digit discrimination task). The emogradCPT consists of digits that gradually fade from one to the next every 800ms, with participants responding to most digits (90% of trials) and withholding responses to rare digits (10% of trials). The task is associated with substantial and stable individual differences, with performance correlating significantly with network connectivity both during task performance and in resting states. The emogradCPT task is an important new paradigm in attention research, providing insights into the neural network of sustained attention.

OTHER OUTCOMES:
Hamilton Depression Scale | Weeks 1, 2, 3, 4, and 5
  The Hamilton Depression Scale (HAM-D) is a clinician-administered 17-item questionnaire assessing the severity of depressive symptoms. Each item measures a depressive symptom (e.g., feelings of guilt, anxiety somatic). Items are rated on a 5-point (0 to 4) or 3-point (0 to 2) scale.
Generalized Anxiety Disorder-7 | Weeks 1, 2, 3, 4, and 5
  The Generalized Anxiety Disorder-7 (GAD-7) assesses anxiety symptom severity over the past two weeks with seven items rated from 0 (not at all) to 3 (nearly every day). An additional item assesses how difficult these symptoms have made functioning, which is rated from "not difficult at all" to "extremely difficult." Total scores use items 1-7 and range from 0 to 21. A score of 10 or greater represents a cut point for identifying cases of GAD, and cut points of 5, 10, and 15 could be interpreted as representing mild, moderate, and severe levels of anxiety.
Pittsburgh Sleep Quality Index | Weeks 1, 2, 3, 4, and 5
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report questionnaire assessing sleep quality in clinical populations. It has seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The PSQI has both Likert-type and open-ended questions. Scores for the ordinal questions range from 0 to 3, with higher scores indicating more acute sleep disturbances.
Patient-rated Inventory of Side-Effects | Weeks 1, 2, 3, 4, and 5
  The Patient-rated Inventory of Side Effects (PRISE) is a 32-item self-report questionnaire assessing the presence and severity of side effects experienced by patients from a medication. Each item is rated on a 4-point scale (0 to 3). Items are summed for total scores, and higher scores indicate greater severity and impact of side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- James J. Peters Veterans Affairs Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided